CLINICAL TRIAL: NCT06453590
Title: Palliative Treatment of Distal Malignant Biliary Obstruction by Endoscopic Stents: Uncovered, Partially Covered, or Fully Covered Metal Stents: A Prospective Randomized Multicenter Study
Brief Title: Treatment of Distal Malignant Biliary Obstruction by Uncovered, Partially Covered, or Fully Covered Metal Stents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180436
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Non-resectable; Bile Duct Cancer; Papillary Carcinoma; Duodenal Cancer
Keywords: distal malignant biliary obstruction; ERCP; SEMS; Palliative
MeSH Terms: conditions — Bile Duct Neoplasms; Carcinoma, Papillary; Duodenal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, to either of three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Uncovered SEMS (Experimental): Allocated to treatment with an uncovered SEMS in the distal bile duct.
  Interventions: Procedure: Randomization to uncovered SEMS treating jaundice due to distal malignant biliary obstruction.
- Partially covered SEMS (Experimental): Allocated to treatment with a partially covered SEMS in the distal bile duct.
  Interventions: Procedure: Randomization to partially covered SEMS treating jaundice due to distal malignant biliary obstruction.
- Fully covered SEMS (Experimental): Allocated to treatment with a fully covered SEMS in the distal bile duct.
  Interventions: Procedure: Randomization to fully covered SEMS treating jaundice due to distal malignant biliary obstruction.

INTERVENTIONS:
Procedure: Randomization to uncovered SEMS treating jaundice due to distal malignant biliary obstruction. — Patients with jaundice due to distal malignant biliary obstruction in whom surgical resection is not possible are treated at ERCP with metal stents, SEMS. The study is comparing three types of commercially available SEMS, Patients are randomized and allocated to either of three stent types (SEMS), uncovered, partially covered , or fully covered.
  Arms: Uncovered SEMS
Procedure: Randomization to partially covered SEMS treating jaundice due to distal malignant biliary obstruction. — Patients with jaundice due to distal malignant biliary obstruction in whom surgical resection is not possible are treated at ERCP with metal stents, SEMS. The study is comparing three types of commercially available SEMS, Patients are randomized and allocated to either of three stent types (SEMS), uncovered, partially covered , or fully covered.
  Arms: Partially covered SEMS
Procedure: Randomization to fully covered SEMS treating jaundice due to distal malignant biliary obstruction. — Patients with jaundice due to distal malignant biliary obstruction in whom surgical resection is not possible are treated at ERCP with metal stents, SEMS. The study is comparing three types of commercially available SEMS, Patients are randomized and allocated to either of three stent types (SEMS), uncovered, partially covered , or fully covered.
  Arms: Fully covered SEMS

SUMMARY:
The goal of this randomized controlled trial is to compare uncovered, partially covered, and fully covered self-expandable metal stents (SEMS) in the palliative treatment of distal malignant biliary obstruction in a Swedish multicenter study.

The main questions it aims to answer is: Is the stent patency rate different depending of stent type? Is the stent patency time different depending of stent type? Is the patient survival different between the groups? Which complications are seen, and do they differ between the groups? Are there different mechanisms behind the stent failure depending on stent type?

Patients will at ERCP, with a guidewire passed through the stenosis in the bile duct, be allocated to either uncovered, partially covered, and fully covered (SEMS). Totally, 450 patients will be recruited, 150 in each study arm, according to the power analysis.

Patients will be followed in a monthly surveillance by a study nurse up to 12 months after stent insertion. Endpoints are: alive after 12 months with a patent stent, death with a patent stent, stent dysfunction with a subsequent intervention i.e. repeated ERCP or PTC = "objective stent failure", stent dysfunction, jaundice or cholangitis, but not intervention has been undertaken due to a poor condition of the patient, "clinical stent failure", the patient has undergone curative surgery or a bilio-enteric by-pass (a gastro-enteroanastomosis or a duodenal stent is not a reason for exclusion), the patient refuses further follow-up.

DETAILED DESCRIPTION:
Background

Malignancies causing distal malignant biliary obstruction may arise from the pancreas, distal bile duct, the papilla of Vater or the duodenum. Pancreatic cancer is more common with an incidence of 11.9/100,000/year, the other diagnoses account for 2.5/100,000/year, thus a total incidence of some 14.4/100,000/year.

The above-mentioned tumors may cause occlusion of the bile duct with subsequent jaundice. The liver function is impaired, and itching caused by the jaundice is disturbing. Only 15-20% of patients are suitable for curative surgery since symptoms often are vague, and the diagnoses is delayed. Thus, at presentation the tumor may be locally advanced or metastasized. High age and comorbidity may also make surgery impossible. Therefore, therapy is often palliative not least aiming at relieving the jaundice.

The aim of stent treatment is to relieve the jaundice, and symptoms associated with the bile duct occlusion. The ERCP-technique is in general the first choice in the biliary intervention. The stenting may be complicated by dysfunction of the drainage, which may be caused by stent occlusion by debris or tumor overgrowth/ingrowth, and stent migration is not uncommon. A repeated biliary intervention is needed but may be difficult or even impossible due to tumor progression. Thus, it is important that the stent treatment is effective with a rapid relief of jaundice, and that the patency time is long.

Initially, plastic stents were used in the ERCP procedures, but now self-expandable metal stents (SEMS) are more common. There are several randomized controlled trials (RCTs) including one of our own group, and metanalyses showing that SEMS have a longer patency time, and are more cost-effective than the plastic stents in the treatment of distal malignant biliary obstruction. SEMS were initially made of steel but now nitinol alloys are more commonly used and have been found superior having a longer patency time/less rate of stent failure as demonstrated in a recent study. When first developed SEMS were manufactured without a covering (uncovered, UC-SEMS) but in order to prevent tumor ingrowth through the metal mesh SEMS were developed with a plastic covering, covered, C-SEMS. The covering may include the whole length of the SEMS (fully covered, FC-SEMS) or spare the 0.5-1 cm ends of the SEMS (semicovered, SC-SEMS).

There are several RCTs comparing UC-SEMS to SC-SEMS. Results are conflicting with some RCTs demonstrating that SC-SEMS have a longer patency time whereas other have not detected any difference between the two types of SEMS. FC-SEMS have been introduced more recently with different outcomes as compared to UC-SEMS. There are no RCTs comparing FC-SEMS to SC-SEMS and UC-SEMS.

UC-SEMS will often attach firmly to the tissue in the stricture, but tumor ingrowth may impair stent function. The covering may prevent ingrowth but there is increased risk migration. The bare proximal end of the SC-SEMS may decrease this risk but in analogy to UC-SEMS they may attach firmly and preclude stent exchange. Contrarily, FC-SEMS may be exchanged in case of dysfunction. Apart from tumor ingrowth and stent dislocation SEMS dysfunction may be caused by proximal or distal overgrowth or epithelial hyperplasia on the inside of the stent.

In conclusion, FC-SEMS may have advantages as compared to SC-SEMS or UC-SEMS, but these three stent types have not been compared in RCTs.

Aim

The aim of the study is to investigate which type of SEMS is superior with respect to the rate of stent failure and patency time (primary outcome). Also, the mechanisms behind the stent failures are analyzed. The frequency and types of complications are studied, and the patent survival time is recorded. The study is also exploring if there is a difference in difficulty in the placement of the three types of stents.

Methods

The current study is a Swedish, three-armed randomized controlled multicenter trial enrolling 450 patients. These patients with distal, malignant biliary obstruction are not suitable for a radical resection (advanced/metastasized disease, comorbidity, high age) are palliatively treated with SEMS. Patients have been investigated by multi-phase CT. Palliative oncological therapy may also be used. After oral and written consent, the patients are randomized to receive a single 10 mm in diameter UC-SEMS, SC-SEMS, or FC-SEMS inserted at ERCP with a length of six or eight cm, multiple stenting is not allowed. Randomization is performed at ERCP when the guide wire has passed the stenosis in the bile duct. 150 patients are allocated to each arm using a randomization list and sealed envelopes. Blocks of ten envelopes are distributed to the participating centers and refilled on demand. The study has been approved by the Swedish Ethical Review Authority (2017/416).

If the patient condition improves after stenting or the radiology after reevaluation demonstrates that a resection is possible the patient will leave the study and proceed to surgery. The placement of a SEMS in this situation as a temporary biliary drainage, before a resection, is no disadvantage. Contrarily, with the superior function of a SEMS as compared to a plastic stent a more rapid biliary relief without early stent failure is accomplished without making surgery more difficult. Thus, it is acceptable that occasional patients are included in a palliative setting, and after reevaluation may proceed to surgery.

The statistical calculations have been performed by the Uppsala Clinical Research Center, UCR. According to the power calculation a difference in stent failure of 14% may be detected with a power of 80%, alpha =0.05, if 150 patients are included in each study arm. A smaller difference in not judged to be clinically significant. The inclusion time is estimated to be three years, and the follow-up time is 12 months.

There are thirteen participating hospitals, seven university hospitals, and six other major hospitals. The participating centers are:

University hospital in Uppsala, Karolinska university hospital in Huddinge, University hospital in Örebro, University hospital in Lund, University hospital in Malmö, Sahlgrenska University hospital in Gothenburg, University hospital in Umeå, South hospital in Stockholm, Danderyds hospital in Stockholm, Capio S:t Görans hospital in Stockholm, Skaraborgs hospital in Skövde, Central hospital in Västerås, Central hospital in Karlstad.

Inclusion

1. Obstructive jaundice (S-Bilirubin > 50 μmol /L). Initial treatment according to the local routine, laboratory test, abdominal CT, often a thoracic CT, and US. These investigations along with the clinical information support the finding of a distal malignant occlusion, and an ERCP is performed.
2. The ERCP demonstrates a seemingly malignant distal biliary stenosis located more than 2 cm below the hilum of the liver.
3. The patient has been found not suitable for curative surgery having a locally to advanced tumor (not a candidate for down-staging) or metastatic decease. The patient age and comorbidity may also preclude major surgery. If the investigations and evaluation is not complete at the time of the ERCP it is permitted to place a temporary plastic endoprosthesis.
4. Patient information. The study has been approved by the Swedish Ethical Review Authority (2017/416) as a multicenter study including an approval for all of the participating centers. The approval of the patient may be withdrawn during the course of the study and will not affect the further treatment which is carried out according to the routine of the participating clinic.
5. Randomization. If the patient has agreed to participate in the study the randomization is performed at the ERCP procedure when the biliary tract has been cannulated, and the guide wire has passed the stenosis. The patient is allocated to UC SEMS, SC, or FC SEMS by the method of sealed, opaque envelopes.

Endpoint of follow-up -12 months - is when/if:

1. The patient has been followed >12 months with a patent stent.
2. The patient expires with a patent stent <12 months.
3. The patient has been found resectable and undergone curative surgery or a bilio-enteric by-pass (a gastro-enteroanastomosis or a duodenal stent is not a reason for exclusion).
4. Stent dysfunction with a subsequent intervention i.e. repeated ERCP or PTC = "objective stent failure".
5. Stent dysfunction, jaundice or cholangitis, but not intervention has been undertaken due to a poor condition of the patient, "clinical stent failure" is also an endpoint.
6. The patient refuses further follow-up.

Follow-up

There is a follow-up 1 month after the ERCP/randomization including laboratory tests, and if the patient condition permits, also a visit at the out-patient clinic. The following monthly checks are performed by phone with questions regarding symptoms of stent dysfunction.

Significance

If one stent type is superior it should be recommended for further use. If the stents are equal there is an argument for inserting only FC SEMS since they also can be extracted, and replaced when occluded, which may be a better alternative than stent in stent placement (plastic endoprosthesis or SEMS). Parallel to the evolvement of new oncological strategies there will probably be a demand for SEMS extraction or replacement i.e. radio frequency, irreversible electroporation, or photodynamic treatment. Moreover, in a situation when a benign condition cannot be excluded the option of a SEMS removal is important. The storage of SEMS in the endoscopy units will also be simplified, and cheaper if there is only need for one type of SEMS.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 20 years.
* The biliary stenosis located > 2 cm below the hilum of the liver, and with a malignant appearance.
* The patient history, and clinical data supporting a malignant bile duct stenosis.
* S-Bilirubin > 50 μmol/L.
* Curative surgery or down-staging not possible due to an advanced decease, or surgery is precluded by high age or co-morbidity. Temporary placement of a plastic endoprosthesis allowed, and after reevaluation within 4 weeks the patient may enter the study.
* The patient has received oral and written information about the study and accepted to participate.
* CT and/or Ultrasound has been performed.

Exclusion Criteria:

* Informed consent has not been obtained or denied.
* The presence of significant intrahepatic stenoses caused by metastatic disease with also intrahepatic obstruction of the bile flow. A malignant stenosis in the hilum of the liver, or a tumor stricture located < 2cm below the hilum of the liver.
* The patient is probably a candidate for curative surgery or down-staging.
* Suspicion of a benign biliary obstruction.
* Anatomical situation making ERCP impossible i.e. prior surgical interventions or a tumor stenosis of the duodenum. If the ERCP is not successful at the first attempt a repeated procedure or a PTC rendezvouz is allowed within one week.
* Prior biliary drainage (> 4 weeks earlier).
* Increased risk of bleeding (INR >1.5)
* The patient has previously been included in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Stent patency rate | During the follow-up time from insertion of the SEMS (inclusion of the study) until reaching an endpoint (up to 12 months with a patent stent or until stent failure occurs) the rate of patent SEMS in the three different groups is calculated
  Stent patency rate of the three different types of SEMS
Stent patency time | The time, days, of patency of the SEMS during follow-up (up to 12 months) until reaching an endpoint is calculated.
  The time, days, of patency of the SEMS in the three different types of SEMS

SECONDARY OUTCOMES:
Patient survival time | The time, days, of survival after stent insertion (inclusion in the study) until death, or up to 12 months.
  Survival time of patients in the three groups of different SEMS
Mechanisms of stent failure | During the follow-up, from the time of stent insertion until a stent failure is established (up to 12 months), the reason is analyzed at the time of repeated ERCP
  Different reasons of stent failure is analyzed, ingrowth, overgrowth, migration, food impaction.
Adverse events | During follow-up from the time of stent insertion complications are registered until an endpoint is reached (up to 12 months).
  Complications arising after stent insertion, stent failure, cholangitis, pancreatitis, bleeding, perforation, cholecystitis.
Difficulty of stent insertion | This outcome is registered during the ERCP procedure.
  Problems arising at ERCP deploying the SEMS as easy, moderately difficult, or difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Linder, MD, PhD, Principal Investigator — Karolinska university hospital, Karolinska Institutet, Stockholm, Sweden.
Locations (12):
- Sweden (12):
  - Danderyds hospital, Danderyd
  - Sahlgrenska University hospital, Gothenburg
  - Central Hospital Karlstad, Karlstad
  - University Hospital Lund, Lund
  - University Hospital Malmö, Malmo
  - University Hospital Örebro, Örebro
  - Skaraborgs Hospital Skövde, Skövde
  - Capio S:t Görans hospital, Stockholm
  - Stockholm South Hospital, Stockholm
  - University Hospital of Umeå, Umeå
  - University hospital Uppsala, Uppsala
  - Central Hospital Västerås, Västerås

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available.
  Individual participant data that underline the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared.
  Study protocol, statistical analysis plan, consent form, clinical study report, and analytic code will be available.
  Data will be available beginning 9 months and ending 72 months after article publication.
  Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose may get access to the data.
  Individual data used in metaanalyses may be provided.
  We may provide deidentified sets of data which was acquired and analyzed in our statistical program.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Nine months after publication up to 72 months
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose may get access to the data. Individual data used in metaanalyses may be provided.

REFERENCES:
- [Background] Cavell LK, Allen PJ, Vinoya C, Eaton AA, Gonen M, Gerdes H, Mendelsohn RB, D'Angelica MI, Kingham TP, Fong Y, Dematteo R, Jarnagin WR, Kurtz RC, Schattner MA. Biliary self-expandable metal stents do not adversely affect pancreaticoduodenectomy. Am J Gastroenterol. 2013 Jul;108(7):1168-73. doi: 10.1038/ajg.2013.93. Epub 2013 Apr 2. PMID 23545711
- [Background] Chen MY, Lin JW, Zhu HP, Zhang B, Jiang GY, Yan PJ, Cai XJ. Covered Stents versus Uncovered Stents for Unresectable Malignant Biliary Strictures: A Meta-Analysis. Biomed Res Int. 2016;2016:6408067. doi: 10.1155/2016/6408067. Epub 2016 Mar 16. PMID 27051667
- [Background] Cotton PB, Garrow DA, Gallagher J, Romagnuolo J. Risk factors for complications after ERCP: a multivariate analysis of 11,497 procedures over 12 years. Gastrointest Endosc. 2009 Jul;70(1):80-8. doi: 10.1016/j.gie.2008.10.039. Epub 2009 Mar 14. PMID 19286178
- [Background] Seaton RA, Nathwani D, Phillips G, Millar R, Davey P. Clinical record keeping in patients receiving antibiotics in hospital. Health Bull (Edinb). 1999 Mar;57(2):128-33. PMID 12811903
- [Background] Gardner TB, Spangler CC, Byanova KL, Ripple GH, Rockacy MJ, Levenick JM, Smith KD, Colacchio TA, Barth RJ, Zaki BI, Tsapakos MJ, Gordon SR. Cost-effectiveness and clinical efficacy of biliary stents in patients undergoing neoadjuvant therapy for pancreatic adenocarcinoma in a randomized controlled trial. Gastrointest Endosc. 2016 Sep;84(3):460-6. doi: 10.1016/j.gie.2016.02.047. Epub 2016 Mar 10. PMID 26972022
- [Background] Irisawa A, Katanuma A, Itoi T. Otaru consensus on biliary stenting for unresectable distal malignant biliary obstruction. Dig Endosc. 2013 May;25 Suppl 2:52-7. doi: 10.1111/den.12069. PMID 23617650
- [Background] Isayama H, Komatsu Y, Tsujino T, Sasahira N, Hirano K, Toda N, Nakai Y, Yamamoto N, Tada M, Yoshida H, Shiratori Y, Kawabe T, Omata M. A prospective randomised study of "covered" versus "uncovered" diamond stents for the management of distal malignant biliary obstruction. Gut. 2004 May;53(5):729-34. doi: 10.1136/gut.2003.018945. PMID 15082593
- [Background] Isayama H, Mukai T, Itoi T, Maetani I, Nakai Y, Kawakami H, Yasuda I, Maguchi H, Ryozawa S, Hanada K, Hasebe O, Ito K, Kawamoto H, Mochizuki H, Igarashi Y, Irisawa A, Sasaki T, Togawa O, Hara T, Kamada H, Toda N, Kogure H. Comparison of partially covered nitinol stents with partially covered stainless stents as a historical control in a multicenter study of distal malignant biliary obstruction: the WATCH study. Gastrointest Endosc. 2012 Jul;76(1):84-92. doi: 10.1016/j.gie.2012.02.039. Epub 2012 Apr 5. PMID 22482918
- [Background] Itoi T, Sofuni A, Itokawa F, Tonozuka R, Ishii K. Current status and issues regarding biliary stenting in unresectable biliary obstruction. Dig Endosc. 2013 May;25 Suppl 2:63-70. doi: 10.1111/den.12062. PMID 23617652
- [Background] Kim HS, Lee DK, Kim HG, Park JJ, Park SH, Kim JH, Yoo BM, Roe IH, Moon YS, Myung SJ. Features of malignant biliary obstruction affecting the patency of metallic stents: a multicenter study. Gastrointest Endosc. 2002 Mar;55(3):359-65. doi: 10.1067/mge.2002.121603. PMID 11868009
- [Background] Kitano M, Yamashita Y, Tanaka K, Konishi H, Yazumi S, Nakai Y, Nishiyama O, Uehara H, Mitoro A, Sanuki T, Takaoka M, Koshitani T, Arisaka Y, Shiba M, Hoki N, Sato H, Sasaki Y, Sato M, Hasegawa K, Kawabata H, Okabe Y, Mukai H. Covered self-expandable metal stents with an anti-migration system improve patency duration without increased complications compared with uncovered stents for distal biliary obstruction caused by pancreatic carcinoma: a randomized multicenter trial. Am J Gastroenterol. 2013 Nov;108(11):1713-22. doi: 10.1038/ajg.2013.305. Epub 2013 Sep 17. PMID 24042190
- [Background] Kullman E, Frozanpor F, Soderlund C, Linder S, Sandstrom P, Lindhoff-Larsson A, Toth E, Lindell G, Jonas E, Freedman J, Ljungman M, Rudberg C, Ohlin B, Zacharias R, Leijonmarck CE, Teder K, Ringman A, Persson G, Gozen M, Eriksson O. Covered versus uncovered self-expandable nitinol stents in the palliative treatment of malignant distal biliary obstruction: results from a randomized, multicenter study. Gastrointest Endosc. 2010 Nov;72(5):915-23. doi: 10.1016/j.gie.2010.07.036. PMID 21034892
- [Background] Lee JH, Krishna SG, Singh A, Ladha HS, Slack RS, Ramireddy S, Raju GS, Davila M, Ross WA. Comparison of the utility of covered metal stents versus uncovered metal stents in the management of malignant biliary strictures in 749 patients. Gastrointest Endosc. 2013 Aug;78(2):312-24. doi: 10.1016/j.gie.2013.02.032. Epub 2013 Apr 13. PMID 23591331
- [Background] Linder S, Bostrom L, Nilsson B. Pancreatic cancer in sweden 1980-2000: a population-based study of hospitalized patients concerning time trends in curative surgery and other interventional therapies. J Gastrointest Surg. 2006 May;10(5):672-8. doi: 10.1016/j.gassur.2005.10.005. PMID 16713540
- [Background] Linder S, Bostrom L, Nilsson B. Pancreatic carcinoma incidence and survival in Sweden in 1980-2000: a population-based study of 16,758 hospitalized patients with special reference to different therapies. Eur J Surg Oncol. 2007 Jun;33(5):616-22. doi: 10.1016/j.ejso.2006.12.022. Epub 2007 Feb 20. PMID 17317081
- [Background] Luigiano C, Ferrara F, Cennamo V, Fabbri C, Bassi M, Ghersi S, Consolo P, Morace C, Polifemo AM, Billi P, Ceroni L, Alibrandi A, D'Imperio N. A comparison of uncovered metal stents for the palliation of patients with malignant biliary obstruction: nitinol vs. stainless steel. Dig Liver Dis. 2012 Feb;44(2):128-33. doi: 10.1016/j.dld.2011.08.015. Epub 2011 Sep 15. PMID 21924691
- [Background] Moss AC, Morris E, Mac Mathuna P. Palliative biliary stents for obstructing pancreatic carcinoma. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD004200. doi: 10.1002/14651858.CD004200.pub4. PMID 16625598
- [Background] Zorron Pu L, de Moura EG, Bernardo WM, Baracat FI, Mendonca EQ, Kondo A, Luz GO, Furuya Junior CK, Artifon EL. Endoscopic stenting for inoperable malignant biliary obstruction: A systematic review and meta-analysis. World J Gastroenterol. 2015 Dec 21;21(47):13374-85. doi: 10.3748/wjg.v21.i47.13374. PMID 26715823
- [Background] Saleem A, Leggett CL, Murad MH, Baron TH. Meta-analysis of randomized trials comparing the patency of covered and uncovered self-expandable metal stents for palliation of distal malignant bile duct obstruction. Gastrointest Endosc. 2011 Aug;74(2):321-327.e1-3. doi: 10.1016/j.gie.2011.03.1249. Epub 2011 Jun 17. PMID 21683354
- [Background] Saxena P, Diehl DL, Kumbhari V, Shieh F, Buscaglia JM, Sze W, Kapoor S, Komanduri S, Nasr J, Shin EJ, Singh V, Lennon AM, Kalloo AN, Khashab MA. A US Multicenter Study of Safety and Efficacy of Fully Covered Self-Expandable Metallic Stents in Benign Extrahepatic Biliary Strictures. Dig Dis Sci. 2015 Nov;60(11):3442-8. doi: 10.1007/s10620-015-3653-5. Epub 2015 Apr 8. PMID 25850628
- [Background] Song TJ, Lee JH, Lee SS, Jang JW, Kim JW, Ok TJ, Oh DW, Park DH, Seo DW, Lee SK, Kim MH, Kim SC, Kim CN, Yun SC. Metal versus plastic stents for drainage of malignant biliary obstruction before primary surgical resection. Gastrointest Endosc. 2016 Nov;84(5):814-821. doi: 10.1016/j.gie.2016.04.018. Epub 2016 Apr 22. PMID 27109456
- [Background] Soderlund C, Linder S. Covered metal versus plastic stents for malignant common bile duct stenosis: a prospective, randomized, controlled trial. Gastrointest Endosc. 2006 Jun;63(7):986-95. doi: 10.1016/j.gie.2005.11.052. PMID 16733114
- [Background] Soderlund C, Linder S, Bergenzaun PE, Grape T, Hakansson HO, Kilander A, Lindell G, Ljungman M, Ohlin B, Nielsen J, Rudberg C, Stotzer PO, Svartholm E, Toth E, Frozanpor F. Nitinol versus steel partially covered self-expandable metal stent for malignant distal biliary obstruction: a randomized trial. Endoscopy. 2014 Nov;46(11):941-8. doi: 10.1055/s-0034-1377936. Epub 2014 Oct 16. PMID 25321620
- [Background] Telford JJ, Carr-Locke DL, Baron TH, Poneros JM, Bounds BC, Kelsey PB, Schapiro RH, Huang CS, Lichtenstein DR, Jacobson BC, Saltzman JR, Thompson CC, Forcione DG, Gostout CJ, Brugge WR. A randomized trial comparing uncovered and partially covered self-expandable metal stents in the palliation of distal malignant biliary obstruction. Gastrointest Endosc. 2010 Nov;72(5):907-14. doi: 10.1016/j.gie.2010.08.021. PMID 21034891
- [Background] Ung KA, Stotzer PO, Nilsson A, Gustavsson ML, Johnsson E. Covered and uncovered self-expandable metallic Hanarostents are equally efficacious in the drainage of extrahepatic malignant strictures. Results of a double-blind randomized study. Scand J Gastroenterol. 2013 Apr;48(4):459-65. doi: 10.3109/00365521.2012.758766. Epub 2013 Feb 4. PMID 23373541
- [Background] Walter D, van Boeckel PG, Groenen MJ, Weusten BL, Witteman BJ, Tan G, Brink MA, Nicolai J, Tan AC, Alderliesten J, Venneman NG, Laleman W, Jansen JM, Bodelier A, Wolters FL, van der Waaij LA, Breumelhof R, Peters FT, Scheffer RC, Leenders M, Hirdes MM, Steyerberg EW, Vleggaar FP, Siersema PD. Cost Efficacy of Metal Stents for Palliation of Extrahepatic Bile Duct Obstruction in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):130-8. doi: 10.1053/j.gastro.2015.03.012. Epub 2015 Mar 17. PMID 25790742
- [Background] Yang MJ, Kim JH, Yoo BM, Hwang JC, Yoo JH, Lee KS, Kang JK, Kim SS, Lim SG, Shin SJ, Cheong JY, Lee KM, Lee KJ, Cho SW. Partially covered versus uncovered self-expandable nitinol stents with anti-migration properties for the palliation of malignant distal biliary obstruction: A randomized controlled trial. Scand J Gastroenterol. 2015;50(12):1490-9. doi: 10.3109/00365521.2015.1057219. Epub 2015 Jul 1. PMID 26133200
- [Background] Jang S, Stevens T, Parsi MA, Bhatt A, Kichler A, Vargo JJ. Superiority of Self-Expandable Metallic Stents Over Plastic Stents in Treatment of Malignant Distal Biliary Strictures. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e182-e195. doi: 10.1016/j.cgh.2020.12.020. Epub 2020 Dec 18. PMID 33346140
- [Background] Yamashita Y, Tachikawa A, Shimokawa T, Yamazaki H, Itonaga M, Sakai Y, Sugiyama H, Nakai Y, Tanaka K, Isayama H, Kitano M. Covered versus uncovered metal stent for endoscopic drainage of a malignant distal biliary obstruction: Meta-analysis. Dig Endosc. 2022 Jul;34(5):938-951. doi: 10.1111/den.14260. Epub 2022 Mar 17. PMID 35114036
- [Background] Suksai N, Kamalaporn P, Chirnaksorn S, Siriyotha S. Factors associated with patency of self-expandable metal stents in malignant biliary obstruction. BMC Gastroenterol. 2023 Nov 14;23(1):392. doi: 10.1186/s12876-023-03028-3. PMID 37964198
- [Background] Yamao K, Takenaka M, Ogura T, Hashimoto H, Matsumoto H, Yamamoto M, Ikeura T, Kurita A, Li ZL, Shiomi H, Chiba Y, Kudo M, Sanuki T. Utility and Safety of a Novel Fully Covered Metal Stent in Unresectable Distal Malignant Biliary Obstruction. Dig Dis Sci. 2020 Dec;65(12):3702-3709. doi: 10.1007/s10620-020-06114-8. Epub 2020 Feb 8. PMID 32036515
- [Background] Ghazi R, AbiMansour JP, Mahmoud T, Martin JA, Law RJ, Levy MJ, Abu Dayyeh BK, Storm AC, Petersen BT, Chandrasekhara V. Uncovered versus fully covered self-expandable metal stents for the management of distal malignant biliary obstruction. Gastrointest Endosc. 2023 Oct;98(4):577-584.e4. doi: 10.1016/j.gie.2023.05.047. Epub 2023 May 16. PMID 37201725
- [Background] Vanella G, Coluccio C, Cucchetti A, Leone R, Dell'Anna G, Giuffrida P, Abbatiello C, Binda C, Fabbri C, Arcidiacono PG. Fully covered versus partially covered self-expandable metal stents for palliation of distal malignant biliary obstruction: a systematic review and meta-analysis. Gastrointest Endosc. 2024 Mar;99(3):314-322.e19. doi: 10.1016/j.gie.2023.10.023. Epub 2023 Oct 7. PMID 37813199
- [Background] Tamura T, Yamai T, Uza N, Yamasaki T, Masuda A, Tomooka F, Maruyama H, Shigekawa M, Ogura T, Kuriyama K, Asada M, Matsumoto H, Takenaka M, Mandai K, Osaki Y, Matsumoto K, Sanuki T, Shiomi H, Yamagata Y, Doi T, Inatomi O, Nakanishi F, Emori T, Shimatani M, Asai S, Fujigaki S, Shimokawa T, Kitano M. Adverse events of self-expandable metal stent placement for malignant distal biliary obstruction: a large multicenter study. Gastrointest Endosc. 2024 Jan;99(1):61-72.e8. doi: 10.1016/j.gie.2023.08.004. Epub 2023 Aug 19. PMID 37598864
- See also: Link to details about cancer incidence i Sweden — https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/dokument-webb/statistik/cancer-i-siffror-2023.pdf